CLINICAL TRIAL: NCT06237608
Title: Acceptability and Feasibility of an Adapted DBT-informed Skills Group for Gender Diverse Young People Co-delivered in a Charity Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Gendered Intelligence (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DBTGI24
Record Dates: First submitted 2024-01-11; First posted 2024-02-01 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2024-03

CONDITIONS: Emotional Regulation
Keywords: emotional regulation; gender diverse
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: 16-week LGBTQ+ -adapted DBT skills group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): Attend DBT-informed skills group intervention
  Interventions: Behavioral: Dialectical behavioural therapy (DBT)-informed skills group

INTERVENTIONS:
Behavioral: Dialectical behavioural therapy (DBT)-informed skills group — 16 week 1.5hr DBT-informed skills group facilitated by the lead researcher and two charity facilitators

SUMMARY:
Gender diverse (e.g. trans or non-binary) young people are at higher risk of self-harm and may be more likely to access support through gender-diverse-specific 3rd sector charities. Dialectical behavioural therapy (DBT) is a transdiagnostic intervention targeting emotion dysregulation, self-harm and suicidality and is recommended by best-practice clinical guidelines; There is developing evidence that DBT skills training can be offered as an effective stand-alone intervention.The current study, therefore, aims to evaluate the feasibility, acceptability and early indicators of effectiveness of a DBT-informed skills group intervention in a gender diverse charity setting. The intervention will be co-facilitated with a gender-diverse support worker from the charity to develop the therapeutic skills of the charity staff working with the young people, whilst they provide specialist knowledge and valuable lived experience.

Research questions

1. Is the intervention feasible to deliver in a charity setting?
2. Is the intervention acceptable to participants and charity facilitators?

Participants will attend a 16-week group intervention. They will complete questionnaire to assess acceptability at the end of the intervention. Attrition rates, training time, and questionnaires will be used to assess feasibility. Outcome measures will also be completed by the participants every three weeks to indicate possible effectiveness of the intervention. The outcomes will include emotion dysregulation, coping skills, anxiety, depression and suicidal behaviours.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-25 years old
* Identify as gender diverse
* Receiving support from Gendered Intelligence
* Support worker identified and self-report emotion regulation difficulties.

Exclusion Criteria:

* In acute crisis at point of recruitment and start of the intervention such as active suicidal ideation with active plans, or severe self-harm requiring intensive interventions such as inpatient or crisis care.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Identify as gender diverse- Gender diversity refers to the representation of people whose gender identity does not conform to socially defined norms. This includes (but is not restricted to) transgender people (whose gender identity does not correspond with their assigned sex at birth) and non-binary people (whose gender identity does not fit within the gender binary of male or female).
Enrollment: 12 (Actual)
Dates: Start 2024-02-03 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of intervention | 16 weeks
  1. Short, bespoke feedback questionnaire completed at the end of each session regarding content and delivery.
Acceptability of intervention | 16 weeks
  2. Client Satisfaction Questionnaire will be completed post-intervention.
Feasibility of intervention | 16 weeks
  1. Eligibility rates at screening
Feasibility of intervention | 16 weeks
  2. Attrition rates at each stage of recruitment - initial number of participants identified by Gendered Intelligence, number of participants approached, number of participants who consented to discuss the project with the researcher, number of participants who consented to take part, number of participants who completed treatment.
Feasibility of intervention | 16 weeks
  3. Attendance and completion rates of the intervention 4. Cost and time to train a charity support worker 5. Number of clinician hours to deliver the intervention and outcome monitoring 6. Number of hours from charity to deliver the intervention 7. How feasible the intervention was to attend (via self-report questionnaire) 8. How feasible the intervention was to deliver (via self-report questionnaire completed by the co-facilitators)
Feasibility of intervention | 16 weeks
  4. Cost and time to train a charity support worker
Feasibility of intervention | 16 weeks
  5. Number of clinician hours to deliver the intervention and outcome monitoring 6. Number of hours from charity to deliver the intervention 7. How feasible the intervention was to attend (via self-report questionnaire) 8. How feasible the intervention was to deliver (via self-report questionnaire completed by the co-facilitators)
Feasibility of intervention | 16 weeks
  6. Number of hours from charity to deliver the intervention
Feasibility of intervention | 16 weeks
  7. How feasible the intervention was to attend (via self-report questionnaire) 8. How feasible the intervention was to deliver (via self-report questionnaire completed by the co-facilitators)
Feasibility of intervention | 16 weeks
  8. How feasible the intervention was to deliver (via self-report questionnaire completed by the co-facilitators)

SECONDARY OUTCOMES:
Emotion dysregulation | Every 2 weeks for 4 weeks, and then every three weeks for 16 weeks once the intervention begins.
  The Difficulties in Emotion Regulation Scale. Higher scores indicate more severe emotion dysregulation difficulties.
Use of DBT coping skills | Every 2 weeks for 4 weeks, and then every three weeks for 16 weeks once the intervention begins.
  The DBT Ways of Coping Checklist
Anxiety | Every 2 weeks for 4 weeks, and then again after 16 weeks.
  Generalised Anxiety Disorder Assessment. Higher scores indicate higher levels of anxiety.
Depression | Every 2 weeks for 4 weeks, and then again after 16 weeks.
  Patient Health Questionnaire. Higher scores indicate higher levels of depression.
Internalised transphobia | Every 2 weeks for 4 weeks, and then every three weeks for 16 weeks once the intervention begins.
  Gender Minority Stress and Resilience Measure. Higher scores indicate higher internalised transphobia.
Gender-related negative future expectations | Every 2 weeks for 4 weeks, and then again after 16 weeks.
  Gender Minority Stress and Resilience Measure. Higher scores indicate higher gender-related negative future expectations.
Gender-related community connectedness | Every 2 weeks for 4 weeks, and then every three weeks for 16 weeks once the intervention begins.
  Gender Minority Stress and Resilience Measure. Higher scores indicate higher gender-related community connectedness.
Gender-specific pride | Every 2 weeks for 4 weeks, and then every three weeks for 16 weeks once the intervention begins.
  Gender Minority Stress and Resilience Measure. Higher scores indicate higher gender-specific pride
Suicidal behaviours | Every 2 weeks for 4 weeks, and then every three weeks for 16 weeks once the intervention begins.
  Frequencies of self-harm, suicidal behaviours, A&E attendances, and inpatient bed days.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Stock, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No